CLINICAL TRIAL: NCT04953442
Title: Fit 24: Using Technology to Improve Activity and Sleep in Hispanic Youth
Brief Title: Fit 24 Technology Intervention YOUTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Erica Gabrielle Soltero Ngwolo, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-49195
Record Dates: First submitted 2021-06-02; First posted 2021-07-08 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Fitbit Device Self-Determination Theory Text Messages
  Interventions: Behavioral: Fit 24
- Wait List Control (No Intervention): Informational flyer of evidence-based strategies on engaging in healthy physical activity and sleep lifestyle habits.

INTERVENTIONS:
Behavioral: Fit 24 — This 12-week goal-setting intervention will test the feasibility of using a Fitbit watch and motivational text messaging to improve physical activity and sleep in Hispanic youth (14-16 years of age) with obesity. Youth will be prompted to set weekly steps per day and hours of sleep per night goals. Text messages will be grounded in the Self-Determination Theory and will provide evidence-based strategies, support, and motivation to encourage youth to meet their goals.
  Arms: Intervention

SUMMARY:
The purpose of this study is to examine the effects of a goal-setting intervention that utilizes a Fitbit device and text messaging to improve physical activity and sleep in Hispanic adolescents with obesity.

DETAILED DESCRIPTION:
Hispanic adolescents are disproportionately burdened by obesity and type 2 diabetes compared to non-Hispanic white youth. Disparities in T2D emerge early in life and are driven in part by unhealthy lifestyle behaviors including low levels of physical activity, excessive time spent in sedentary behaviors and short sleep durations. Given that Hispanic youth are the fastest growing pediatric subgroup in the U.S., developing strategies to promote healthy lifestyle behaviors and addressing T2D disparities is a public health imperative. Wearable activity monitoring devices like Fitbits are designed to continuously monitor both wake time and sleep behaviors. Therefore the purpose of this study is to examine the feasibility, acceptability, and preliminary efficacy of a 12-week technology-based intervention that uses a Fitbit and text messages grounded in the Self-Determination Theory to promote healthy lifestyle habits and reduce risk for type 2 diabetes among a Hispanic adolescents with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Self identify as Hispanic or Latino
* obese, defined as body mass index percentile (BMI%) ≥ 95th percentile
* Ages of 14-16 years
* Own his or her own cellphone.

Exclusion Criteria:

* Taking a medication(Steroids) or diagnosed with a condition (i.e. sleep (i.e. sleep apnea) that influences activity, sleep, and/or cognition
* Recent hospitalization or injury that prevents normal physical activity
* pregnant
* currently enrolled in an exercise program or currently using a personal activity monitoring device like Fitbit.

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-04-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soltero EG, Lopez C, Musaad SM, O'Connor TM, Thompson D. Fit24, a digital health intervention to reduce type 2 diabetes risk among Hispanic youth: Protocol for a feasibility pilot study. Contemp Clin Trials. 2023 Apr;127:107117. doi: 10.1016/j.cct.2023.107117. Epub 2023 Feb 10. PMID 36775009
- [Derived] Soltero EG, Lopez C, Hernandez E, O'Connor TM, Thompson D. Technology-Based Obesity Prevention Interventions Among Hispanic Adolescents in the United States: Scoping Review. JMIR Pediatr Parent. 2022 Nov 4;5(4):e39261. doi: 10.2196/39261. PMID 36331547

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Youth were recruited from local pediatric clinics, community-based organizations (eg, Houston Public Library and Baker Ripley Community Developers), and by word of mouth. Interested participants were screened via telephone for eligibility criteria.
Pre-assignment Details: After baeline data collection participating youth were randomized (1:1 randomization) to the intervention or to a waitlist control group. The youth in the intervention received a Fitbit Charge 5 device and daily SMS text messages grounded in SDT. Youth randomized to the waitlist control group received a Fitbit Charge 5 device and a one-page informational handout on PA and sleep guidelines.
Groups:
- Wait List Control: Youth randomized to the waitlist control group received a Fitbit Charge 5 device and a one-page informational handout on PA and sleep guidelines.
- Intervention: The youth in the intervention received a Fitbit Charge 5 device and daily SMS text messages grounded in SDT.
Period: Overall Study
Arm/Group | Wait List Control | Intervention
Started | 21 | 22
Completed | 18 | 22
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Wait List Control | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] — Age was self-reported.
  years | 15.09 (0.768) | 14.95 (0.95) | 15.02 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex was self-reported as sex assigned at birth. Population: Sex was self-reported as sex assigned at birth.
  Participants
    Female | 14 | 13 | 27
    Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Self Reported demographic survey completed by parents Population: Self Reported demographic survey completed by parents
  Participants
    Hispanic or Latino | 22 | 21 | 43
    Not Hispanic or Latino | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number Participants Recruited
Description: We will record the number participants recruited, screened, and enrolled in the study.
Time Frame: 4 months
Population: This is the count of participants that were enrolled in each intervention arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Wait List Control | Intervention
Number analyzed (Participants) | 21 | 22
Participants | 21 | 22

2. Primary Outcome: Number of Technical Issues Experienced by Participants
Description: We will record the number of technical issues experienced by participants throughout the study.
Time Frame: 12-weeks
Measure: Number; unit: number of technical issues
Arm/Group | Wait List Control | Intervention
Number analyzed (Participants) | 21 | 22
number of technical issues | 0 | 16

3. Primary Outcome: Percentage of Participants That Are Satisfied With Participation in the Study
Description: We will use a survey to assess the % of participants that are satisfied with participation in the study.
Time Frame: 12-weeks
Population: Only participants originally randomized to the intervention completed the exit survey to indicate their satisfaction with the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Wait List Control | Intervention
Number analyzed (Participants) | 0 | 22
Participants | 0 | 19

4. Secondary Outcome: Average Minutes of Physical Activity
Description: Physical activity was measured using accelerometry for a 7 day protocol.
Time Frame: Baseline and 12-weeks post intervention
Reporting Status: Not Posted, anticipated posting 2025-09

5. Other Pre Specified Outcome: Average of Minutes of Sleep Per Night
Description: Sleep will be assessed using accelerometry to assess average minutes/night using a 24-hour, 7-day accelerometer protocol.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: minutes/night
Arm/Group | Intervention | Wait List Control
Number analyzed (Participants) | 22 | 21
minutes/night | 503.3 (87.7) | 470.98 (60.54)

6. Other Pre Specified Outcome: Body Mass Index
Description: Height and weight will be measured to the nearest 0.1cm and 0.1 kg, using a portable stadiometer and research scale to calculate BMI percentile.
Time Frame: 4 months
Reporting Status: Not Posted, anticipated posting 2025-09

7. Other Pre Specified Outcome: Psychological Need Fulfillment as Assessed Using Psychological Need Satisfaction in Exercise Scale (PNSE)
Description: The Psychological Need Satisfaction in Exercise Scale (18-items) will be used to assess psychological needs fulfillment. The total possible scores in the PNSE are 6-108 with higher scores reflect greater perceptions of psychological need fulfillment.
Time Frame: 4 months
Reporting Status: Not Posted, anticipated posting 2025-09

8. Other Pre Specified Outcome: Autonomous Motivation for Physical Activity as Assessed Using Behavioural Regulation in Exercise Questionnaire-2 (BREQ-2)
Description: The Behavioural Regulation in Exercise Questionnaire-2 (23-items) will be used to assess autonomous motivation for physical activity. The total possible scores on the BREQ-2 are -24 to 24, with a higher score indicating reflect more self-determined motivation whereas negative scores indicate less self-determined motivation.
Time Frame: 4 months
Reporting Status: Not Posted, anticipated posting 2025-09

ADVERSE EVENTS:
Time Frame: From enrollment up to 14 weeks
Description: Given that no adverse events were experienced, there is no relevant information about adverse event collection.
Arm/Group | Intervention | Wait List Control
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 0/22 | 0/21

LIMITATIONS AND CAVEATS:
Limitations included issues related to the feasibility of the Fitbit device. Several participants reported that the Fitbit watch band was uncomfortable and irritated their skin. The Fitbit device syncs through the Fitbit app once a Bluetooth connection has been established; however, sync issues occurred in this study due to a loss of Bluetooth connection, differences in app settings, or differences in operating systems that did not allow for the automatic or continuous syncing of the device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT04953442/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT04953442/SAP_001.pdf